CLINICAL TRIAL: NCT03364101
Title: The Poweroff Study
Brief Title: The Poweroff Sleep Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-01020
Record Dates: First submitted 2017-11-21; First posted 2017-12-06 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PowerOff (Experimental): PowerOff is a nutraceutical and a blend of nine ingredients for sleep, including: melatonin; California Poppy; L-Cystine; Glycine; and Magnolia Officinalis
  Interventions: Dietary Supplement: POWEROFF Capsule
- Placebo (Placebo Comparator): The placebo pill will be manufactured at the same facility and appear identical in all aspects. However, the control agent will feature non-active ingredients with regards to sleep.Capsules will be instructed to commence on day 7 of the study after baseline appointment
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Placebo Capsule — Composition of the placebo is 100% organic rice flour, manufactured at a facility New York State licensed to produce pharmaceuticals. Capsules will be instructed to commence on day 7 of the study after baseline appointment.
  Arms: Placebo
Dietary Supplement: POWEROFF Capsule — blend of California Poppy Aerial Part Extract, L-Cystine, L-Theanine,GABA (proprietary Phosphatidylcholine-Palmitic Acid-Oleic Acid Complex), 5-HTP, Magnolia Officinalis Bark Extract, Glycine, Melatonin with 0.5mg of Vitamin B6 (as pyridoxal-5-phosphate).
  Arms: PowerOff

SUMMARY:
The primary objective is to explore the relationship between experimental condition (placebo or PowerOff) and sleep quality between pre-study and post-study. In addition, volunteers will wear actigraphy watches that collect objective measures of sleep, such as total sleep time, and these data points will be compared pre- and post-study.

ELIGIBILITY:
Inclusion Criteria:

* Sleep/Wake History. Participants must currently maintain a regular sleep/wake schedule (±2 hr average bedtime) and express willingness to continue to follow a regular sleep-wake schedule.
* Drug/Alcohol Use. Participants must be drug-free (including nicotine). No medications (prescription or over the counter) that significantly affect circadian rhythms or sleep are allowed. Subjects must report no history of drug or alcohol dependency to be included in the study.
* Evaluation of Medical Suitability. Only healthy men and women are to be selected for this study. Subjects will be free from any acute, chronic, or debilitating medical conditions. Normality will be established on the basis of self-report clinical history and diagnoses/. Any subject with symptoms of active illness, such as fever, infection, or hypertension, will be excluded.
* Evaluation of Psychiatric/Psychological Suitability. Individuals with a history of psychiatric illnesses or psychiatric disorders will be excluded. Individuals who are unaware of specific psychiatric diagnoses but had a history of treatment with antidepressant, neuroleptic medications, or major tranquilizers will be excluded from the study. Subjects will also be questioned to demonstrate their full understanding of the requirements, demands, and risks of the study and informed of the option to withdraw at any time.

Exclusion Criteria:

* Older adults are known to experience decreased depth of non-rapid eye movement sleep (NREM), as well as lesser amounts of deep sleep (NREM3), They therefore spend greater amounts of their sleep time in less protected lighter sleep stages. For these reasons, older adults (above age 65) will be excluded from the study.
* Individuals whom have had a negative or paradoxical response to an OTC sleep supplement or OTC sleep medication (Nyquil zzz's, Benadryl, melatonin, valerian, etc.).
* Individuals who are or are planning to become pregnant in the next 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Change in score on Pittsburgh Sleep Quality Index (PSQI) | 12 Days
  measures quality and pattern of sleep in adults. It differentiates "poor" from "good" sleep quality

SECONDARY OUTCOMES:
Sleep Duration | 12 Days
  collected objectively via the sleep monitoring actigraphy wristwatch
Sleep Duration | 12 Days
  collected subjectively using self-reported questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States